CLINICAL TRIAL: NCT05325294
Title: Evaluation of the Advanced Hybrid Closed Loop (AHCL) System in Type 1 Adult and Pediatric Subjects Utilizing Lyumjev® Insulin Lispro-aabc
Brief Title: Evaluation of the Advanced Hybrid Closed Loop (AHCL) System in Type 1 Adults and Pediatrics Utilizing Lyumjev®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP335
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- MiniMed 780G System Utilizing Insulin Lyumjev® (Experimental): Subjects with insulin-requiring type 1 diabetes age 7-80 using the MiniMed 780G system with Insulin Lyumjev® for a period of three months.
  Interventions: Device: MiniMed 780G System

INTERVENTIONS:
Device: MiniMed 780G System — MiniMed™ 780G Insulin Pump, Guardian™ 4 Glucose Sensor, and Guardian 4 Transmitter; used with Insulin Lyumjev® insulin lispro-aabc

SUMMARY:
This US study will evaluate the safety and effectiveness of utilizing insulin Lyumjev® lispro-aabc in the MiniMed™ 780G System in Type 1 adult and pediatric subjects in a home setting to support product and system labeling.

DETAILED DESCRIPTION:
This study is a multi-center, single arm study in insulin-requiring adult and pediatric subjects with type 1 diabetes on the MiniMed™ 780G system using Lyumjev® insulin lispro-aabc and Medtronic Extended infusion set and reservoir. The run-in period and study period will be approximately 120 days long.

A total of up to 250 subjects with insulin-requiring type 1 diabetes age 7-80 will be enrolled at up to 25 investigational centers across the United States in order to have at least 200 subjects enter the study period. Up to 125 subjects will be enrolled in the pediatric age group (7-17 years of age) and up to 125 in the adult age group (18 years or older).

ELIGIBILITY:
Inclusion Criteria:

1. Age 7-80 years at time of screening.
2. Has a clinical diagnosis of type 1 diabetes:

   1. 14-80 years of age: A clinical diagnosis of type 1 diabetes for 2 years or more as determined via medical record or source documentation by an individual qualified to make a medical diagnosis.
   2. 7-13 years of age: A clinical diagnosis of type 1 diabetes for 1 year or more as determined via medical record or source documentation by an individual qualified to make a medical diagnosis.
3. Does not require a legally authorized representative to consent on their behalf due to mental or intellectual disability.
4. Subject or parent/caregiver is literate and able to read the language offered in the pump or pump materials.
5. Subject and/or legally authorized representative is willing to provide informed consent for participation.
6. Is willing to perform fingerstick blood glucose measurements as needed.
7. Is willing to wear the system continuously throughout the study.
8. Must have a minimum daily insulin requirement (Total Daily Dose) of greater than or equal to 8 units and a maximum total daily dose of 250 units or less.
9. Has a Glycosylated hemoglobin (HbA1c) less than 10% (as processed by Central Lab) at time of screening visit.

   Note: All HbA1c blood specimens will be sent to and tested by a National Glycohemoglobin Standardization Program (NGSP) certified Central Laboratory. HbA1c testing must follow NGSP standards.
10. Has thyroid-stimulating hormone (TSH) in the normal range OR if the TSH is out of normal reference range, the Free T3 is below or within the lab's reference range and Free T4 is within the normal reference range.
11. Uses pump therapy for greater than 6 months (with or without CGM experience) prior to screening
12. Is willing to upload data from the study pump, must have Internet access, and a computer system, or compatible smartphone that meets the requirements for uploading the study pump.
13. Is willing to take one of the following insulins and can financially support the use of insulin preparations as required during the run-in period:

    1. Humalog (insulin lispro injection)
    2. NovoLog (insulin aspart injection)
    3. Admelog(insulin lispro injection)
14. Is willing to take Lyumjev insulin during the study period (supplied via Sponsor).

Exclusion Criteria:

1. Has hypersensitivity to insulin lispro or one of the excipients in Lyumjev®
2. Has a history of 2 or more episodes of severe hypoglycemia, which resulted in any the following during the 6 months prior to screening:

   1. Medical assistance (i.e., Paramedics, Emergency Room [ER] or Hospitalization)
   2. Coma
   3. Seizures
3. Has been hospitalized or has visited the ER in the 6 months prior to screening resulting in a primary diagnosis of uncontrolled diabetes.
4. Has had DKA in the last 6 months prior to screening visit.
5. Will not tolerate tape adhesive in the area of sensor placement as assessed by a qualified individual.
6. Has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection).
7. Is female of child-bearing potential and result of pregnancy test is positive at screening.
8. Is sexually active female of child-bearing potential and is not using a form of contraception deemed reliable by the investigator.
9. Is female and plans to become pregnant during the course of the study
10. Is being treated for hyperthyroidism at time of screening.
11. Has diagnosis of adrenal insufficiency.
12. Has taken any oral, injectable, or intravenous (IV) glucocorticoids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV glucocorticoid during the course of the study.
13. Is using hydroxyurea at time of screening or plans to use it during the study.
14. Is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks.
15. Is currently abusing illicit drugs.
16. Is currently abusing marijuana.
17. Is currently abusing prescription drugs.
18. Is currently abusing alcohol.
19. Using pramlintide (Symlin), DPP-4 inhibitor, liraglutide (Victoza or other GLP-1 agonists), metformin, canagliflozin (Invokana or other SGLT2 inhibitors) at time of screening.
20. Has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator.
21. Has elective surgery planned that requires general anesthesia during the course of the study.
22. Has sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening.
23. Plans to receive red blood cell transfusion or erythropoietin over the course of study participation.
24. Is diagnosed with current eating disorder such as anorexia or bulimia.
25. Has been diagnosed with chronic kidney disease that results in chronic anemia.
26. Has a hematocrit that is below the normal reference range of lab used.
27. Is on dialysis.
28. Has serum creatinine of >2 mg/dL.
29. Has celiac disease that is not adequately treated as determined by the investigator.
30. Has had any of the following cardiovascular events within 1 year of screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, or ventricular rhythm disturbances.
31. Has had history of cardiovascular event 1 year or more from the time of screening without

    1. a normal EKG and stress test within 6 months prior to screening or during screening or
    2. clearance from a qualified physician prior to receiving the study devices if there is an abnormal EKG or stress test.
32. Has 3 or more cardiovascular risk factors listed below without a normal EKG within 6 months prior to screening or during screening or clearance from a qualified physician if there is an abnormal EKG:

    * Age >35 years
    * Type 1 diabetes of >15 years' duration
    * Presence of any additional risk factor for coronary artery disease
    * Presence of microvascular disease (proliferative retinopathy or nephropathy, including microalbuminuria)
    * Presence of peripheral vascular disease
    * Presence of autonomic neuropathy
33. Is a member of the research staff involved with the study.
34. Has used a MiniMed 780G pump prior to screening

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Stanford University, Palo Alto, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Barbara Davis Center, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - East Coast Institute for Research (Memorial Hospital), Jacksonville, Florida
  - University of South Florida Diabetes Center, Tampa, Florida
  - Atlanta Diabetes, Atlanta, Georgia
  - East Coast Institute for Research - Macon, Macon, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Rocky Mountain, Idaho Falls, Idaho
  - Barry J Reiner MD LLC, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - International Diabetes Center, Saint Louis Park, Minnesota
  - The Docs LLC, Las Vegas, Nevada
  - Physicians East, Greenville, North Carolina
  - Texas Diabetes, Austin, Texas
  - Diabetes and Glandular Disease Clinic, P.A, San Antonio, Texas
  - Rainier Research, Renton, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 244 subjects (120 with age 7-17 and 124 with age 18-80) enrolled at the beginning, with 23 (12 with age 7-17 and 11 with age 18-80) screen failure, 10 subjects (7 with age 7-17 and 3 with age 18-80) early withdrawn prior the study period, 211 subjects (101 with age 7-17 and 110 with age 18-80) started the study and became the Intention to Treat Population.
Groups:
- Subjects 7-17 Years of Age: Subjects with insulin-requiring type 1 diabetes age 7-17 using the MiniMed 780G system with Insulin Lyumjev® for a period of three months.
  MiniMed 780G System: MiniMed™ 780G Insulin Pump, Guardian™ 4 Glucose Sensor, and Guardian 4 Transmitter; used with Insulin Lyumjev® insulin lispro-aabc
- Subjects 18-80 Years of Age: Subjects with insulin-requiring type 1 diabetes age 18-80 using the MiniMed 780G system with Insulin Lyumjev® for a period of three months.
  MiniMed 780G System: MiniMed™ 780G Insulin Pump, Guardian™ 4 Glucose Sensor, and Guardian 4 Transmitter; used with Insulin Lyumjev® insulin lispro-aabc
Period: Overall Study
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age
Started | 101 | 110
Completed | 97 | 101
Not Completed | 4 | 9
Not completed — Adverse Event | 3 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Sponsor Request | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intention to Treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age | Total
Number analyzed (Participants) | 101 | 110 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.0 (2.6) | 45.0 (14.2) | 29.7 (19.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 49 | 100
  Male | 50 | 61 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 7 | 26
  Not Hispanic or Latino | 81 | 103 | 184
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 8 | 4 | 12
  White | 85 | 103 | 188
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 4 | 2 | 6
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.0 (4.6) | 28.8 (5.3) | 25.6 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint - Change in HbA1c
Description: The overall mean change in HbA1c from baseline to end of 3-month study period. Non-inferiority test.
Time Frame: 3 months
Population: Intention to Treat Population with available data. Two subjects aged 7-17 and two subject aged 18-80 did not collect A1C at the end of the study period, so 99 subjects aged 7-17 and 108 subjects aged 18-80 were analyzed at end of study period and the change from baseline to end of study period.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age
Number analyzed (Participants) | 99 | 108
percentage of HbA1c | -0.1 (0.7) | -0.4 (0.6)
Statistical Analysis 1: Comparison: Subjects 7-17 Years of Age; Test type: Non-Inferiority — The overall mean change in HbA1c from baseline to end of 3-month study period. The mean change will be estimated and compared to a threshold of -0.38% with a margin of 0.4%; p = 0.133, t-test, 1 sided; Mean difference from baseline to exit = -0.1, 95% CI 2-sided [-0.2 to 0.1] — This is one arm study, the differences of HbA1c from baseline to exit were summarized for this endpoint
Statistical Analysis 2: Comparison: Subjects 18-80 Years of Age; Test type: Non-Inferiority — The overall mean change in HbA1c from baseline to end of 3-month study period. The mean change will be estimated and compared to a threshold of -0.5% with a margin of 0.4%; p < 0.001, Wilcoxon (Mann-Whitney); Mean difference from baseline to exit = -0.4, 95% CI 2-sided [-0.6 to -0.3] — This is one arm study, the differences of HbA1c from baseline to exit were summarized for this endpoint

2. Primary Outcome: Primary Effectiveness Endpoint - Percent of Time in Range (TIR 70-180 mg/dL)
Description: The mean % of time in range (TIR 70-180 mg/dL). Non-inferiority test.
Time Frame: Last 6-7 weeks of 3 month study period
Population: Intention to Treat Population with available data. Three subjects aged 7-17 and eight subject aged 18-80 did not have enough SG points at the last 6 weeks of the study period, so 98 subjects aged 7-17 and 102 subjects aged 18-80 were analyzed at last 6 weeks of study period.
Measure: Mean (Standard Deviation); unit: percentage of Time in Range (TIR 70-180
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age
Number analyzed (Participants) | 98 | 102
percentage of Time in Range (TIR 70-180 | 68.6 (10.3) | 77.6 (9.6)
Statistical Analysis 1: Comparison: Subjects 7-17 Years of Age; Test type: Non-Inferiority — The mean % of time in range (TIR 70-180 mg/dL) will be estimated and compared to a threshold of 65.3% with a margin of -7.5% and a significance level of 0.025 (one-sided); p < 0.001, t-test, 1 sided; Mean of Final Value = 68.6, 95% CI 2-sided [66.6 to 70.7] — This is one arm study, the Percent of Time in Range (TIR70-180 mg/dL) from the last 6-7 weeks of 3 month study period was summarized for this endpoint
Statistical Analysis 2: Comparison: Subjects 18-80 Years of Age; Test type: Non-Inferiority — The mean % of time in range (TIR 70-180 mg/dL) will be estimated and compared to a threshold of 73.7% with a margin of -7.5% and a significance level of 0.025 (one-sided); p < 0.001, t-test, 1 sided; Mean of Final Value = 77.6, 95% CI 2-sided [75.7 to 79.4] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Secondary Effectiveness Endpoint 1 - Percent of Time in Hypoglycemia (< 54 mg/dL)
Description: The mean % of time in hypoglycemia (< 54 mg/dL). Non-inferiority test.
Time Frame: Last 6-7 weeks of 3 month study period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of Time in Hypoglycemia (< 54
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age
Number analyzed (Participants) | 98 | 102
percentage of Time in Hypoglycemia (< 54 | 0.4 (0.5) | 0.2 (0.3)
Statistical Analysis 1: Comparison: Subjects 7-17 Years of Age; Test type: Non-Inferiority — The mean % of time in hypoglycemia (< 54 mg/dL) will be estimated and compared to a threshold of 0.71% with a margin of 2% and a significance level of 0.025 (one-sided); p < 0.001, Wilcoxon (Mann-Whitney); Mean of Final Value = 0.4, 95% CI 2-sided [0.3 to 0.5] — This is one arm study, the Percent of Time in Hypoglycemia (< 54 mg/dL) from the last 6-7 weeks of 3 month study period was summarized for this endpoint
Statistical Analysis 2: Comparison: Subjects 18-80 Years of Age; Test type: Non-Inferiority — The mean % of time in hypoglycemia (< 54 mg/dL) will be estimated and compared to a threshold of 0.86% with a margin of 2% and a significance level of 0.025 (one-sided); p < 0.001, Wilcoxon (Mann-Whitney); Mean of Final Value = 0.2, 95% CI 2-sided [0.2 to 0.3] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Secondary Effectiveness Endpoint 2 - Percent of Time in Range (TIR 70-180 mg/dL)
Description: The mean % of time in range (TIR 70-180 mg/dL). Superiority test.
Time Frame: Last 6-7 weeks of 3 month study period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of Time in Range (TIR 70-180
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age
Number analyzed (Participants) | 98 | 102
percentage of Time in Range (TIR 70-180 | 68.6 (10.3) | 77.6 (9.6)
Statistical Analysis 1: Comparison: Subjects 7-17 Years of Age; Test type: Superiority — The mean % of time in range (TIR 70-180 mg/dL) will be estimated and compared to a threshold of 65.3% and a significance level of 0.025 (one-sided); p < 0.001, t-test, 1 sided; Mean of Final Value = 68.6, 95% CI 2-sided [66.6 to 70.7] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Subjects 18-80 Years of Age; Test type: Superiority — The mean % of time in range (TIR 70-180 mg/dL) will be estimated and compared to a threshold of 73.7% and a significance level of 0.025 (one-sided); p < 0.001, t-test, 1 sided; Mean of Final Value = 77.6, 95% CI 2-sided [75.7 to 79.4] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: 3-month Study Period
Description: Only Adverse Events during the study period were posted
Groups:
- Subjects 7-17 Years of Age Study Period: Subjects with insulin-requiring type 1 diabetes age 7-17 using the MiniMed 780G system with Insulin Lyumjev® for a period of three months.
  MiniMed 780G System: MiniMed™ 780G Insulin Pump, Guardian™ 4 Glucose Sensor, and Guardian 4 Transmitter; used with Insulin Lyumjev® insulin lispro-aabc
- Subjects 18-80 Years of Age Study Period: Subjects with insulin-requiring type 1 diabetes age 18-80 using the MiniMed 780G system with Insulin Lyumjev® for a period of three months.
  MiniMed 780G System: MiniMed™ 780G Insulin Pump, Guardian™ 4 Glucose Sensor, and Guardian 4 Transmitter; used with Insulin Lyumjev® insulin lispro-aabc
Arm/Group | Subjects 7-17 Years of Age Study Period | Subjects 18-80 Years of Age Study Period
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/110
Other Adverse Events (participants affected / at risk) | 50/101 | 47/110
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects 7-17 Years of Age Study Period (N=101) | Subjects 18-80 Years of Age Study Period (N=110)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Binocular eye movement disorder (Eye disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Noninfective gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Infusion site bruising (General disorders) | 0 (0) | 1 (1)
Infusion site reaction (General disorders) | 1 (1) | 0 (0)
Infusion site swelling (General disorders) | 1 (2) | 0 (0)
Medical device site dermatitis (General disorders) | 0 (0) | 1 (1)
Medical device site haemorrhage (General disorders) | 1 (1) | 0 (0)
Medical device site irritation (General disorders) | 2 (3) | 2 (2)
Medical device site papule (General disorders) | 0 (0) | 1 (1)
Medical device site reaction (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Physical deconditioning (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 9 (9)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 2 (2)
Infusion site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (6) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 2 (2) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 4 (4)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 10 (11) | 5 (6)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 10 (14) | 11 (18)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (8) | 1 (1)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT05325294/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT05325294/SAP_001.pdf